CLINICAL TRIAL: NCT01551641
Title: A Phase II Clinical Trial on VEGF Expression Interfered by Thalidomide Combined With Concurrent Chemoradiotherapy in Esophageal Cancer
Brief Title: Phase II Trial of Thalidomide Combined With Concurrent Chemoradiotherapy in Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changzhou No.2 People's Hospital (Other)
Responsible Party: Principal Investigator, Suping Sun, Director, Head of Radiation oncology, Principal Investigator, Clinical Professor, Changzhou No.2 People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CZEY-THA-001
Record Dates: First submitted 2012-02-24; First posted 2012-03-13 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Chemoradiotherapy; VEGF; Thalidomide
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Chemoradiotherapy; Thalidomide

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VEGF decressed (Experimental): patients will receive concurrent chemoradiotherapy only
  Interventions: Other: chemoradiotherapy
- thalidomide (Experimental): patients will be given thalidomide concurrent chemoradiotherapy
  Interventions: Drug: thalidomide
- without thalidomide (Experimental): patients will receive concurrent chemoradiotherapy only
  Interventions: Other: without thalidomide

INTERVENTIONS:
Other: chemoradiotherapy — Patients only receive concurrent chemoradiotherapy if their serum VEGF level decrease.
  Other Names: chemo-radiotherapy
  Arms: VEGF decressed
Drug: thalidomide — Patients will be given thalidomide combined with concurrent chemoradiotherapy if their serum VEGF level increase or unchanged.
  Other Names: neurosedyn
  Arms: thalidomide
Other: without thalidomide — Patients only receive concurrent chemoradiotherapy if their serum VEGF level increase or unchanged
  Other Names: without neurosedyn
  Arms: without thalidomide

SUMMARY:
The purpose of this study is to down-regulate VEGF expression in esophageal cancer patients by thalidomide, so to improve their chemoradiotherapy effect. Patients with esophageal cancer receiving chemoradiotherapy were divided into different sub-group according to dynamic change of their VEGF level,and those showed increased or unchanged VEGF were added thalidomide at random. Efficacy and side effect of thalidomide combined with chemoradiotherapy were evaluated, and at the same time, activity of thalidomide on esophageal cancer and its clinical safely were assessed.

DETAILED DESCRIPTION:
Radiotherapy:Patients will be conducted CT simulation, and three-dimensional conformal radiation therapy (3DCRT) was performed. 1.8-2.0 Gy/fraction, 5 fractions a week, with a total dose of 60-72Gy will be delivered for all patients by 6-MV-X-ray of linear accelerator.

Chemotherapy: Patients will be concurrently administered with irradiation every 4 weeks with PT regimen (cis-platinum of 25 mg/m2/d, d1-4; PTX(paclitaxel)of 135mg/m2/d, d1) for 4 cycles. For the first 2-cycles of chemotherapy they will be concurrently given with irradiation and the remained 2 cycles, after irradiation.

Administration of thalidomide: Determine serum VEGF level of the esophageal cancer patients 3-4 weeks after the beginning of radiotherapy, those whose VEGF level, compared with that before radiotherapy, increased or unchanged will be divided into two groups: one is given thalidomide concurrent with the following chemoradiotherapy, 100mg/d at bedtime for the initial week, and if no moderate above side effect occurred 200mg/d from the next week till the end of chemoradiotherapy; the other received concurrent chemoradiotherapy only.

VEGF determination: Peripheral venous blood samples will be taken in one week before, 3-4 weeks during, and in one week after radiotherapy respectively. The serum VEGF will be determined by the double antibody sandwich ELISA.

ELIGIBILITY:
Inclusion Criteria:

* cytologically or histologically confirmed esophageal carcinoma
* age of 20 -80
* Karnofsky performance status ≥ 70
* no treatments prior to enrollment
* at least one measurable lesion on CT, MRI or esophageal barium exam
* normal functions of heart, lung, liver, kidney and bone marrow
* blood exams qualified for chemotherapy, which included hemoglobulin ≥9 g/dl, neutrophil ≥1.5×109/L and platelet (PLT) ≥100×109/L, creatinine ≤1.5 UNL
* informed consent signed

Exclusion Criteria:

* prior treatments of chemotherapy or irradiation
* poor bone marrow, liver and kidney functions, which would make chemotherapy intolerable
* contraindication for irradiation: complete obstruction of esophagus, deep esophageal ulcer, fistula to mediastinum, or haematemesis
* participating in other clinical trials
* pregnancy, breast feeding, or not adopting birth control
* drug or alcohol addiction, uncontrolled epileptic seizure, or psychotic with no ability of self control
* coexisted morbidities that investigators believed not suitable for chemoradiation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-01; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Treatment efficacy | 3 months after completion of treatment
  Treatment efficacy were evaluated by the indexes as Locoregional tumor response. Locoregional tumor response will be evaluated 3 months after completion of treatment according to Response Evaluation Criteria in Solid Tumors (RECIST).

SECONDARY OUTCOMES:
Overall survival (OS) | 1 year and 3 years after completion of treatment
  Overall survival (OS) will be evaluated 1 year and 3 years after completion of treatment using Kaplan-Meier model.
Local progression-free survival (LPFS) | 1 year and 3 years after completion of treatment
  1 year and 3 years after completion of treatment using Kaplan-Meier model.
Safety | 1 week after completion of treatment
  All patients are to be estimated Quality Of Life(such as dizzy, somnolence, queasiness and vomit,anaphylaxis incidence) ,acute radiation reactions such as acute radiation esophagitis and tracheitis incidence(evaluated by the Radiation Therapy Oncology Group (RTOG) toxicity criteria),complete blood cell count(such as leukocyte, neutrophil,hemoglobulin, platelet level), serum biochemistry(such as creatinine level).

CONTACTS AND LOCATIONS:
Overall Officials: Sun Suping, M.D.,PhD., Principal Investigator — Changzhou No.2 People's Hospital
Locations (1):
- Changzhou No.2 People's Hospital, Changzhou, Jiangsu, China